CLINICAL TRIAL: NCT06714084
Title: Cadonilimab in Neoadjuvant Chemotherapy and Maintenance Therapy for Newly Diagnosed, High-risk, Locally Advanced Cervical Cancer :a Multi-center, Prospective, Single-arm Study(CNCMT)
Brief Title: CNCMT：a Multi-center, Prospective, Single-arm Study
Acronym: CNCMT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Collaborators: Yichang Central People's Hospital (Other); Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Principal Investigator, YI HUANG, Archiater, Hubei Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNCMT; ChiCTR2400088236 (Other: chinese clinical trial registry)
Record Dates: First submitted 2024-11-21; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Locally Advanced Cervical Cancer; PD1; CTLA4
Keywords: cervical cancer; Cadonilimab; maintenance therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Neoadjuvant Therapy; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Experimental): Cadonilimab in neoadjuvant chemotherapy and maintenance therapy for newly diagnosed advanced cervical cancer
  Interventions: Drug: Neoadjuvant Chemotherapy (NACT); Drug: maintenance therapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy (NACT) — Two cycles of carbonilumab plus TP regimen neoadjuvant chemotherapy will be implemented to patients with advanced cervical cancer
Drug: maintenance therapy — one years of maintenance therapy with carbonilumab alone will be implemented to patients with advanced cervical cancer receiving standard concurrent chemoradiotherapy

SUMMARY:
To evaluate the safety and efficacy of Cadonilimab in neoadjuvant chemotherapy and maintenance therapy for high-risk advanced cervical cancer receiving concurrent chemoradiotherapy

DETAILED DESCRIPTION:
Cadonilimab is a humanized, bispecific antibody targeting PD-1 and CTLA-4.Studies have verified the efficacy of cadonilimab in recurrent uterine cervical cancer, yet the regiment and the safety and efficacy of cadonilimab in newly diagnosed advanced cervical cancer are still unclear. This study tried to explore the safety and efficacy of cadonilimab in neoadjuvant chemotherapy and maintenance therapy in high-risk advanced cervical cancer receiving concurrent chemoradiotherapy .

Inclusion criteria:

1. Written informed consent must be provided and recorded at the trial site before any trial procedure is initiated;
2. Female patients aged ≥ 18 years and < 75 years;
3. Histologically confirmed diagnosis of cervical malignancy, and the histological type include squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma, and other histological types;
4. Have not received systematic or local anti-tumor treatment for cervical cancer before the first medication, including but not limited to radiotherapy, chemotherapy, immunotherapy, biologics, small molecule targeted therapy, etc;
5. Patients who agree to receive radical synchronous radiotherapy and chemotherapy, and whose researchers have determined that there are no absolute contraindications to radiotherapy and chemotherapy;
6. High risk cervical cancer patients, including those with local cervical tumors>5cm, lymph node metastasis or stage IV patients;
7. The subjects agree to collect tumor tissue and peripheral blood samples required during the screening period and research process, and apply them to relevant studies;
8. Has good organ function;
9. No history of using immune checkpoint inhibitors;
10. Female subjects with fertility must undergo a urine or serum pregnancy test (if the urine pregnancy test result cannot be confirmed as negative, a serum pregnancy test must be performed, based on the serum pregnancy result) within 3 days before the first use of medication, and the result must be negative. If a female subject with fertility has sexual intercourse with an unsterilized male partner, the subject must self screen and adopt an acceptable contraceptive method, and must agree to continue using the contraceptive method for 120 days after the last use of the study drug; Whether to stop contraception after this point in time should be discussed with the researchers. Periodic abstinence and safe period contraception are unacceptable contraceptive methods;
11. Women with fertility refer to those who have not undergone surgical sterilization (i.e. bilateral tubal ligation, bilateral oophorectomy, or total hysterectomy) or have not reached menopause (menopause is defined as a period of at least 12 consecutive months without alternative medical reasons, and serum follicle stimulating hormone levels are within the laboratory reference range for postmenopausal women);
12. Efficient contraceptive methods refer to contraceptive methods with a low failure rate (such as less than 1% per year) when used consistently and correctly. Not all contraceptive methods are efficient. In addition to barrier contraception, female subjects with fertility must also use hormone contraception alone (such as birth control pills) to ensure that pregnancy does not occur
13. ECOG score ≤ 1;
14. Expected survival period>12 weeks;
15. Understand the experimental process and have the ability to comply with the experimental protocol during the duration of the experiment, including cooperating with any treatments, examinations, tests, follow-up, and survey questionnaires required to complete the experiment;
16. The patient is willing to cooperate in completing the quality of life questionnaire survey during the trial treatment and follow-up process, and agrees that the results of these questionnaire surveys will be used for clinical research;

Exclusion criteria:

1. Personnel involved in the development or implementation of research plans;
2. Previously received PD-1/PD-L1 and CTLA-4 bispecific antibody therapy or drugs that synergistically inhibit T cell receptors (such as OX-40, CD137);
3. Individuals who are known to be allergic to the active ingredients or excipients of the investigational drug Cardenimumab;
4. Symptomatic or uncontrolled brain metastases that require simultaneous treatment, including but not limited to surgery, radiation, and/or corticosteroids, or clinical manifestations of spinal cord compression;
5. Currently participating in interventional clinical research treatment, or having received other research drugs or used research instruments for treatment within 4 weeks before the first administration;
6. Diagnosed with other malignant diseases other than cervical cancer within 5 years before the first administration (excluding curative basal cell carcinoma, squamous cell carcinoma of the skin, and/or carcinoma in situ that has undergone curative resection);
7. Within 2 years prior to the first administration, there has been an active autoimmune disease requiring systemic treatment (such as the use of disease relieving drugs, corticosteroids, or immunosuppressants). Alternative therapies (such as thyroid hormone, insulin, or physiological glucocorticoids used for adrenal or pituitary insufficiency) are not considered systemic treatments; Note: Patients with cataracts, Graves' disease, or psoriasis who do not require systematic treatment (within the past 2 years) are not excluded;
8. Within 3 months prior to the first administration, there is active hemoptysis (at least 2.5ml or 1/2 teaspoon of blood is expelled at a time);
9. Receive a live vaccine within one month before the first administration;
10. Note: It is allowed to receive inactivated vaccine for seasonal influenza within 30 days before the first administration; However, intranasal administration of attenuated live influenza vaccine is not allowed.
11. Received platelet or red blood cell transfusion within 4 weeks before the first administration;
12. Have undergone major surgical treatment within 4 weeks prior to the first administration (excluding surgery for biopsy purposes) or are expected to undergo major surgery during the study period;
13. Within 2 weeks before the first administration, he has received systematic systemic treatment with traditional Chinese patent medicines and simple preparations with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural effusion); 14. Within 7 days prior to the first administration, the individual is receiving systemic corticosteroid therapy (excluding topical corticosteroids via nasal spray, inhalation, or other routes) or any other form of immunosuppressive therapy (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor drugs);

15. Note: Physiological doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent) are allowed to be used; 16. Undertook minor surgeries (outpatient/inpatient surgeries requiring local anesthesia, including central venous catheterization) within 48 hours prior to the initial receipt of the study drug; 17. Patients with clinically uncontrollable pleural/peritoneal effusion (those who do not require drainage or have no significant increase in effusion after stopping drainage for 3 days can be enrolled); 18. Severe unhealed wounds, ulcers, or fractures; 19. Known allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation; 20. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive); 21. Active hepatitis B without treatment; 22. Women who are pregnant or breastfeeding, or planning to become pregnant during the study treatment period; 23. There are unresolved previous treatment toxicities in clinical practice (≥ grade 2, excluding hair loss, neuralgia, lymphopenia, and depigmentation of the skin); 24. The presence of any serious or uncontrollable systemic disease; 25. Medical history or disease evidence that may interfere with the trial results, hinder the full participation of the subjects in the study, abnormal treatment or laboratory test values, or other situations that the researchers consider unsuitable for inclusion. The researchers believe that there are other potential risks that are not suitable for participation in this study.

ELIGIBILITY:
Inclusion Criteria:1. Written informed consent must be provided and recorded at the trial site before any trial procedure is initiated; 2. Female patients aged ≥ 18 years and < 75 years; 3. Histologically confirmed diagnosis of cervical malignancy, and the histological type include squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma, and other histological types; 4. Have not received systematic or local anti-tumor treatment for cervical cancer before the first medication, including but not limited to radiotherapy, chemotherapy, immunotherapy, biologics, small molecule targeted therapy, etc; 5. Patients who agree to receive radical synchronous radiotherapy and chemotherapy, and whose researchers have determined that there are no absolute contraindications to radiotherapy and chemotherapy; 6. High risk cervical cancer patients, including those with local cervical tumors>5cm, lymph node metastasis or stage IV patients; 7. The subjects agree to collect tumor tissue and peripheral blood samples required during the screening period and research process, and apply them to relevant studies; 8. Has good organ function; 9. No history of using immune checkpoint inhibitors; 10. Female subjects with fertility must undergo a urine or serum pregnancy test (if the urine pregnancy test result cannot be confirmed as negative, a serum pregnancy test must be performed, based on the serum pregnancy result) within 3 days before the first use of medication, and the result must be negative. If a female subject with fertility has sexual intercourse with an unsterilized male partner, the subject must self screen and adopt an acceptable contraceptive method, and must agree to continue using the contraceptive method for 120 days after the last use of the study drug; Whether to stop contraception after this point in time should be discussed with the researchers. Periodic abstinence and safe period contraception are unacceptable contraceptive methods; 11. Women with fertility refer to those who have not undergone surgical sterilization (i.e. bilateral tubal ligation, bilateral oophorectomy, or total hysterectomy) or have not reached menopause (menopause is defined as a period of at least 12 consecutive months without alternative medical reasons, and serum follicle stimulating hormone levels are within the laboratory reference range for postmenopausal women); 12. Efficient contraceptive methods refer to contraceptive methods with a low failure rate (such as less than 1% per year) when used consistently and correctly. Not all contraceptive methods are efficient. In addition to barrier contraception, female subjects with fertility must also use hormone contraception alone (such as birth control pills) to ensure that pregnancy does not occur 13. ECOG score ≤ 1; 14. Expected survival period>12 weeks; 15. Understand the experimental process and have the ability to comply with the experimental protocol during the duration of the experiment, including cooperating with any treatments, examinations, tests, follow-up, and survey questionnaires required to complete the experiment; 16. The patient is willing to cooperate in completing the quality of life questionnaire survey during the trial treatment and follow-up process, and agrees that the results of these questionnaire surveys will be used for clinical research; -

Exclusion Criteria:1. Personnel involved in the development or implementation of research plans; 2. Previously received PD-1/PD-L1 and CTLA-4 bispecific antibody therapy or drugs that synergistically inhibit T cell receptors (such as OX-40, CD137); 3. Individuals who are known to be allergic to the active ingredients or excipients of the investigational drug Cardenimumab; 4. Symptomatic or uncontrolled brain metastases that require simultaneous treatment, including but not limited to surgery, radiation, and/or corticosteroids, or clinical manifestations of spinal cord compression; 5. Currently participating in interventional clinical research treatment, or having received other research drugs or used research instruments for treatment within 4 weeks before the first administration; 6. Diagnosed with other malignant diseases other than cervical cancer within 5 years before the first administration (excluding curative basal cell carcinoma, squamous cell carcinoma of the skin, and/or carcinoma in situ that has undergone curative resection); 7. Within 2 years prior to the first administration, there has been an active autoimmune disease requiring systemic treatment (such as the use of disease relieving drugs, corticosteroids, or immunosuppressants). Alternative therapies (such as thyroid hormone, insulin, or physiological glucocorticoids used for adrenal or pituitary insufficiency) are not considered systemic treatments; Note: Patients with cataracts, Graves' disease, or psoriasis who do not require systematic treatment (within the past 2 years) are not excluded; 8. Within 3 months prior to the first administration, there is active hemoptysis (at least 2.5ml or 1/2 teaspoon of blood is expelled at a time); 9. Receive a live vaccine within one month before the first administration; 10. Note: It is allowed to receive inactivated vaccine for seasonal influenza within 30 days before the first administration; However, intranasal administration of attenuated live influenza vaccine is not allowed.

11. Received platelet or red blood cell transfusion within 4 weeks before the first administration; 12. Have undergone major surgical treatment within 4 weeks prior to the first administration (excluding surgery for biopsy purposes) or are expected to undergo major surgery during the study period; 13. Within 2 weeks before the first administration, he has received systematic systemic treatment with traditional Chinese patent medicines and simple preparations with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural effusion); 14. Within 7 days prior to the first administration, the individual is receiving systemic corticosteroid therapy (excluding topical corticosteroids via nasal spray, inhalation, or other routes) or any other form of immunosuppressive therapy (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor drugs); 15. Note: Physiological doses of glucocorticoids (≤ 10 mg/day of prednisone or equivalent) are allowed to be used; 16. Undertook minor surgeries (outpatient/inpatient surgeries requiring local anesthesia, including central venous catheterization) within 48 hours prior to the initial receipt of the study drug; 17. Patients with clinically uncontrollable pleural/peritoneal effusion (those who do not require drainage or have no significant increase in effusion after stopping drainage for 3 days can be enrolled); 18. Severe unhealed wounds, ulcers, or fractures; 19. Known allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation; 20. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive); 21. Active hepatitis B without treatment; 22. Women who are pregnant or breastfeeding, or planning to become pregnant during the study treatment period; 23. There are unresolved previous treatment toxicities in clinical practice (≥ grade 2, excluding hair loss, neuralgia, lymphopenia, and depigmentation of the skin); 24. The presence of any serious or uncontrollable systemic disease; 25. Medical history or disease evidence that may interfere with the trial results, hinder the full participation of the subjects in the study, abnormal treatment or laboratory test values, or other situations that the researchers consider unsuitable for inclusion. The researchers believe that there are other potential risks that are not suitable for participation in this study.

-

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate at 12 months | up to 12 months
  Progression-free survival rate at 12 months after receiving treatment
Objective response rate(ORR) of neoadjuvant therapy | About 2 months
  Proportion of patients with complete response（CR） and partial response(PR) of the neoadjuvant therapy

SECONDARY OUTCOMES:
mPFS | through study completion, an average of 24 months
  the median time from the date of treatment to the first of either disease progression, relapse or death from any cause
mOS | through study completion, an average of 6 years
  the median time of patients are alive after starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: HUANG YI, Master's degree, Principal Investigator
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Experimental design, basic information of subjects, experimental results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From December 2024 to December 2030
Access Criteria: Healthcare workers, accessed at the following web site:https://www.chictr.org.cn/showproj.html?proj=233028
URL: https://www.chictr.org.cn/showproj.html?proj=233028